CLINICAL TRIAL: NCT01408667
Title: A Phase 2A, Double-blind, Placebo-controlled, Randomized Study to Evaluate the Safety and Efficacy of TRC150094 in Increasing Insulin Sensitivity in Male Patients With Increased Cardiometabolic Risk
Brief Title: Hyperinsulinemic Euglycemic Clamp Protocol
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT/P015/CMR/2010/02_01; 2011-002398-42 (EudraCT Number)
Record Dates: First submitted 2011-07-29; First posted 2011-08-03 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Metabolic Cardiovascular Syndrome
Keywords: insulin sensitivity; cardiometabolic risk; hyperinsulinemic euglycemic clamp
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — TRC150094

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- TRC150094 (Active Comparator)
  Interventions: Drug: TRC150094

INTERVENTIONS:
Drug: TRC150094 — 50 mg Tablets once a day
  Arms: TRC150094
Other: Placebo — Tablets once daily
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the safety and efficacy of TRC150094 in male patients with cardiometabolic risk. Cardiometabolic risk which is the overall risk of cardiovascular disease (CVD) and diabetes resulting from the presence of hypertension, HDL cholesterol, insulin resistance, dysglycemia and visceral obesity.

DETAILED DESCRIPTION:
20 Subjects will be enrolled in Veeda Clinical research,India and another 20 subjects at Amsterdam, the Netherlands. The maximum duration of participation in the study for each subject will be 9.5 weeks including a less than or equal to 4 weeks screening period, 4 weeks of treatment and a 10 days post treatment follow-up evaluation period.

At each study site, 20 subjects will be enrolled. Each subject will attend the study centre in a fasting state, for a screening visit, 2 study visits (one baseline and one end of treatment), 1 intermediate safety visit and 1 post-study follow-up visit (Total 5 visits). The subjects at each site will be randomized to receive TRC150094 or placebo in a ratio of 1:1. 50 mg dose will be administered once daily (morning) under fasting conditions. Dosing will take place daily on Days 1-28. Subjects will arrive at the study centre for screening visit. Physical examination, vital signs, safety biochemistry and laboratory investigations for verification of inclusion/ exclusion criteria will be performed during screening visit. Subjects meeting all the inclusion criteria and none of the exclusion criteria and who have given their informed consent for the study will be asked to come for the study on Day 0 (or day -1 if required). Baseline investigations (including baseline clamp procedure and hepatic MRS) will be done on Day 0 (or day -1). Subjects will receive properly labelled bottle containing either Active treatment or Placebo as per the randomization number of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be considered eligible for entry in the study if they meet all of the following criteria.

  1. Adult male
  2. Age range 30-65 years at screening
  3. Caucasian or Indian ethnicity
  4. Waist circumference ≥ 102 cm for Caucasians and ≥ 90 cm for Indians at screening.
  5. Fasting Serum Insulin ≥ 10 mU/ml at screening
  6. Blood Pressure ≥ 130/85 mmHg at screening (or patients taking medication for hypertension)
  7. Stable weight during 3 months prior to the study (assessed through medical history of the patient)
  8. Drug naive diabetic patients* or patients with impaired fasting glucose i.e > 100 mg/dl or 5.5 mmol/l and < 200 mg/dl or 11.0 mmol/l Diabetic patients who were taking metformin and have undergone washout for at least 4 weeks before Day 0 and are currently on life style modification as a treatment for diabetes will also be allowed in the study
  9. Willingness to give written informed consent (prior to any study-related procedures being performed) and ability to adhere to the study restrictions and assessments schedule.

     * Diabetic patient is defined as a patient with a documented history of type II DM or a documented history of a fasting glucose > 200mg/dl or 11.0 mmol/l or 2x fasting glucose > 126 mg/dl or 6.9 mmol/l (2x =recorded twice).

Exclusion Criteria:

* Subjects will not be considered eligible for entry in the study if they meet one or more of the following criteria.

  1. Medical history, physical examination, vital signs, clinical laboratory tests, 12-lead ECG and Chest X ray (to exclude tuberculosis in India only) with any significant abnormalities, in the opinion of the investigator.
  2. Subjects with any known somatic illness, including neoplasm, endocrine disorder such as cushing's disease, PCOD and uncontrolled hypothyroidism, neurologic disorder, active infection, or recent surgical procedure within 3 months of the study initiation.
  3. Subject currently using medication, which can influence glucose or FFA metabolism such as fibrates, niacin, ACE inhibitors, PPAR agonists, omega 3 fatty acids.
  4. eGFR < 60 mL/min/1.73m2 at screening as evaluated by Modification of Diet in Renal Disease (MDRD) method.
  5. History of angina, Myocardial Infarction (MI) or stroke since last 6 months.
  6. Hypertension with SBP/DBP ≥160/100 mmHg at screening.
  7. ALT or AST ≥ ULN*3 at screening
  8. History or presence of malignancy.
  9. History of recreational drug use within the last 30 days, or regular consumption of greater than 2 units of alcohol/day.
  10. History of allergy to the test drug or any drug chemically similar to the drug under investigation.
  11. Seropositive for Hepatitis B, Hepatitis C or HIV.
  12. Subjects suffering from any psychiatric (acute or chronic) illness.
  13. Intake of any medication except those permitted in this study (see Section 6.6).
  14. Intake of any investigational drug in the period within 3 months prior to the first dose of study drug.
  15. History of significant blood loss due to any reason, including blood donation, in the 12 weeks prior to the first dose of study drug; or the total blood loss in the last 3 months, including for this study, exceeds 450 mL.
  16. History of any bleeding disorder.
  17. Existence of any surgical or medical condition which, in the judgment of the principal investigator, might interfere with the absorption, distribution, metabolism or excretion of the study drug or might be likely to compromise the safety of the subject.
  18. Inability to communicate or co-operate with the investigator because of language problems, poor mental development or impaired cerebral function.
  19. Inability to comply with study requirements.
  20. Positive drugs of abuse test (at screening) and alcohol breath test.
  21. Heavy smokers (who are smoking >15 cigarettes or equivalent per day).

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The safety of TRC150094 once daily dosing for 4 weeks in male patients with increased cardiometabolic risk will be determined. | 1 month
  Safety parameters will include haematology, safety biochemistry, vital signs, ECG and AE check.
The efficacy (in increasing insulin sensitivity) of TRC150094 once daily dosing for 4 weeks in male patients with increased cardiometabolic risk will be determined. | 1 month
  Efficacy assessment will include Insulin Sensitivity to be determined by:
  Rate of Glucose Disposal Suppression of Endogenous Glucose Production Suppression of rate of lipolysis

SECONDARY OUTCOMES:
The effect of TRC150094 on hepatic fat and metabolic parameters will be evaluated. | 1 month
  Early efficacy markers to be explored includes:
  * Hepatic fat by magnetic resonance spectroscopy
  * Lipid parameters
  * Metabolic markers such as adiponectin, IL-6, TNF-alpha, CRP, glucagon, leptin etc.
The ethnic differences for effect of TRC150094 on Insulin sensitivity parameters will be evaluated. | 1 month
  Difference in insulin sensitivity parameters (rate of glucose disposal) between caucasian and Indian populations.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Stroes, MD, PhD, Principal Investigator — Department of Vascular Medicine, AMC
Locations (1):
- Academic Medical Centre,, Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Background] Zambad SP, Munshi S, Dubey A, Gupta R, Busiello RA, Lanni A, Goglia F, Gupta RC, Chauthaiwale V, Dutt C. TRC150094 attenuates progression of nontraditional cardiovascular risk factors associated with obesity and type 2 diabetes in obese ZSF1 rats. Diabetes Metab Syndr Obes. 2011 Jan 6;4:5-16. doi: 10.2147/DMSOTT.S15323. PMID 21448317
- [Background] Cioffi F, Zambad SP, Chhipa L, Senese R, Busiello RA, Tuli D, Munshi S, Moreno M, Lombardi A, Gupta RC, Chauthaiwale V, Dutt C, de Lange P, Silvestri E, Lanni A, Goglia F. TRC150094, a novel functional analog of iodothyronines, reduces adiposity by increasing energy expenditure and fatty acid oxidation in rats receiving a high-fat diet. FASEB J. 2010 Sep;24(9):3451-61. doi: 10.1096/fj.10-157115. Epub 2010 May 7. PMID 20453112
- [Derived] van der Valk F, Hassing C, Visser M, Thakkar P, Mohanan A, Pathak K, Dutt C, Chauthaiwale V, Ackermans M, Nederveen A, Serlie M, Nieuwdorp M, Stroes E. The effect of a diiodothyronine mimetic on insulin sensitivity in male cardiometabolic patients: a double-blind randomized controlled trial. PLoS One. 2014 Feb 21;9(2):e86890. doi: 10.1371/journal.pone.0086890. eCollection 2014. PMID 24586256